CLINICAL TRIAL: NCT03204656
Title: Selective Bronchial Intubation (SBI) at Marie Lannelongue Hospital (HML) : Epidemiology of Expected and Unexpected Difficult Intubations.
Brief Title: Selective Bronchial Intubation (SBI)
Acronym: SBI
Status: Completed | Type: Observational
Sponsor: Centre Chirurgical Marie Lannelongue (Other)
Responsible Party: Sponsor
Other Study IDs: 2016-A02070-51
Record Dates: First submitted 2017-03-22; First posted 2017-07-02 (Actual); Last update posted 2017-07-02 (Actual); Status verified 2017-05

CONDITIONS: Selective Bronchial Tube
Keywords: difficult orotracheal intubation; selective lung intubation; unexpected difficult selective lung intubation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Difficult orotracheal intubation carries a risk of hemodynamic collapse, neurological sequelae secondary to cerebral anoxia or death. Anesthetic scores and predictive indices are used to predict difficulties and avoid complications for usual tracheal intubation. However, existing indices are not adapted to selective bronchial intubations.

The aim of the study is to determine the incidence of unexpected difficult SBI using conventional screening tests. It is a prospective descriptive epidemiological monocentric study comparing two groups of patients (selective vs. non selective intubations).

ELIGIBILITY:
Inclusion Criteria:

* For adult patients : age greater than or equal to 18 years
* Patients with thoracic, cardiac, vascular or plastic surgery

Exclusion Criteria:

* Intubations performed before admission to the operating room or catheterization room;
* Patient whose age is less than 18 years
* Traditional re-intubation at the end of the procedure after a selective lung IOT;
* Selective re-intubation in a patient previously intubated on arrival at the operating theater;
* IOT in other departments of the HML (intensive care, Pulmonary Postoperative Unit (UPOP), bronchoscopy, hospitalization services, Intensive Care Unit (ICU), etc.).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult patients with intubation during surgery in Marie Lannelongue's hospital
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2017-02-20 (Actual); Primary Completion 2017-05-20 (Actual); Study Completion 2017-05-20 (Actual)

PRIMARY OUTCOMES:
Rate of difficult selective bronchial intubation | 1 day
  Rate (percentage)

SECONDARY OUTCOMES:
Predictive factors of difficult selective bronchial intubation | 1 day
  questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Marie Lannelongue, Le Plessis-Robinson, France

IPD SHARING:
Plan to Share IPD: No